CLINICAL TRIAL: NCT05421364
Title: Effects of Intrauterine Administration of Autologous Peripheral Blood Mononuclear Cells (PBMC) on the Endometrial Cells Populations
Brief Title: Effects of Intrauterine Administration of Autologous PBMC on the Endometrial Cells Populations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nadezhda Women's Health Hospital (Other)
Collaborators: Medical diagnostic laboratory ImunoVita (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10/12042022
Record Dates: First submitted 2022-06-06; First posted 2022-06-16 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Female Infertility
Keywords: Peripheral blood mononuclear cells (PBMC); Female infertility; Endometrium; Endometrial cell populations
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Intervention Model Description: Both prior to and following PBMC treatment endometrial biopsies will be obtained on day 7 after LH peak.
  The endometrial samples will be stained immunohistochemically with antibodies against specific endometrial cell types.The endometrial cell composition and the specific cell types quantities will be evaluated by microscopic observation and flowcytometric analysis.
  The cell composition and their quantities will be compared before and after intrauterine administration of PBMC in the endometrial biopsies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Endometrial cell composition (Experimental): The cell composition and their quantities will be compared before and after intrauterine administration of PBMC in the endometrial biopsies.
  Interventions: Biological: Intrauterine administration of autologous peripheral blood mononuclear cells (PBMC)

INTERVENTIONS:
Biological: Intrauterine administration of autologous peripheral blood mononuclear cells (PBMC) — Approximately 9 ml blood from each patient will be collected on the day of the LH peak by peripheral venipuncture using a 21G butterfly catheter affixed via vacutainer to negative pressure receiving tubes (BD vacutainer acid-citrate-dextrose (ACD-A), REF:366645). PBMC will be isolated by density gradient centrifugation in room-temperature centrifuge set to 400 g for 25 min. PBMCs (1x106cells/ml) suspended in RPMI 1640 supplemented with 10% HSA will be incubated in the presence of 10 IU/ml hHCG for 48 h. On day 2 after LH peak, fresh PBMCs (1x107 cells) will be also obtained from the same patients, these fresh PBMCs will be immediately combined with the 2-day cultured PBMC and suspended in PBS (2x107 cells/200µl). This cell suspension will be carefully introduced in the uterine cavity by catheter on day 2 after LH peak.

SUMMARY:
The behaviour of the endometrium during its receptive phase is highly dependent on the endometrial cell type composition. Each cell type has its role in the endometrial preparation for the invading embryo. Alteration in the immune cells dialogue could be the main reason for unsuccessful implantation in certain patients. Immune cell homeostasis is often improved by intrauterine administration of autologous PBMC.

There have been numerous reports on the positive effects of the intrauterine administration of autologous PBMC on the IVF outcomes (embryo implantation and ongoing pregnancy success). However, there is little data on the direct effect of the PBMC administration on the cell composition of the endometrium. This study will focus on the changes in the endometrial cell populations by PBMC treatment that could lead to IVF outcome improvement.

The aim of this project is to analyze the effect of intrauterine administration of autologous PBMC on the endometrial cell populations and on the IVF outcome parameters (implantation and ongoing pregnancy success as IVF outcome variables).

ELIGIBILITY:
Inclusion Criteria:

* Participating in Assisted Reproduction Treatment
* Presenting altered endometrial immune profile
* Having primary infertility
* Having regular menstrual cycles
* Embryo transfer of euploid embryos

Exclusion Criteria:

* Uterine pathologies
* Endometrial Bacterial infections
* Active endometrial inflammation
* Polycystic ovary syndrome
* Presence of auto anti-bodies such as anti-TPO, anti-TG, ACA, APA, ANA, and anti-dsDNA
* Presence of mutations involving the coagulation system such as deficiency of factor XII, Pro C, Pro S
* Cancer diagnostics
* Positive HIV, HCV or HBV tests

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-12-09 (Actual); Primary Completion 2026-01-03 (Estimated); Study Completion 2026-12-09 (Estimated)

PRIMARY OUTCOMES:
Change in the numbers of certain ednometrial cell populations (immune cells, stem cells, senescent cells) from their levels one month prior intrauterine PBMC administration | One month following intrauterine PBMC administration
  Immunohistochemical analysis
Change in the percentages of the immune cells in the endometrial stroma from their levels one month prior intrauterine PBMC administration | One month following intrauterine PBMC administration
  Flowcytometric analysis
Change in the distance between the endometrial immune cells, stem cells and senescent cells in the endometrial stroma from their initial distances one month prior intrauterine PBMC administration | One month following intrauterine PBMC administration
  Spatial analysis with Visual analysis software

SECONDARY OUTCOMES:
Embryo implantation rate | Two weeks following embryo transfer
  Defined as high levels of human chorionic gonadotropin (hCG) in the peripheral blood
Clinical pregnancy rate | Six to 8 weeks of gestation
  Defined as number of gestational sacs with fetal heart beat, shown by ultrasound in gestational week 6 per number of embryo transferred.

CONTACTS AND LOCATIONS:
Locations (2):
- Bulgaria (2):
  - Nadezhda Women's Health Hospital, Sofia, Sofia
  - Medical diagnostic laboratory Imunovita, Sofia

IPD SHARING:
Plan to Share IPD: No